CLINICAL TRIAL: NCT02174315
Title: Contingency Management Treatment of Alcohol Abuse American Indian People
Brief Title: Motivational Incentives for Alcohol Abstinence in American Indian and Native Alaskan Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Michael McDonell, Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 46593-G
Record Dates: First submitted 2014-05-13; First posted 2014-06-25 (Estimated); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism

ARMS (2):
- Contingency Management (Experimental)
  Interventions: Behavioral: Contingency Management
- Non-Contingent Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Contingency Management
  Arms: Contingency Management

SUMMARY:
This study examines the impact of a culturally tailored version of contingency management treatment on alcohol in 400 alcohol dependent American Indians and Alaskan Natives. Participants will be recruited from addiction treatment agencies and throughout the community. Those who complete a 4 week induction period will be randomized to receive 12 weeks of contingency management or a non-contingent control condition. Individuals will then be followed for an additional 3-months to assess the long term efficacy of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Self reported American Indian/Alaskan Native
* Current alcohol dependence
* 5 or more standard drink on 1 or more occasions in the last 30 days
* Ability to read and speak English
* Ability to provide written informed consent

Exclusion Criteria:

* Illicit drug use greater than alcohol use in the last 90 days
* A risk of dangerous alcohol withdrawal
* Any medical or psychiatric condition, such as organic brain disorder, dementia, or psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2014-10-01; Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Change in alcohol use as assessed by ethyl glucuronide detection in urine | Twice weekly for twelve weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael McDonell, PhD, Principal Investigator — Washington State University
Locations (1):
- Contact PI, Pullman, Washington, United States

REFERENCES:
- [Derived] Hirchak KA, Kordas G, Lyons AJ, Herron J, Jansen K, Shaw J, McPherson SM, Roll J, Buchwald D, McDonell MG; HONOR Study Team. Investigating Secondary Alcohol Outcomes in a Contingency Management Intervention among American Indian and Alaska Native Adults. J Addict Med. 2023 May-Jun 01;17(3):e177-e182. doi: 10.1097/ADM.0000000000001116. Epub 2022 Dec 21. PMID 37267179
- [Derived] Hirchak KA, Lyons AJ, Herron JL, Kordas G, Shaw JL, Jansen K, Avey JP, McPherson SM, Donovan D, Roll J, Buchwald D, Ries R, McDonell MG; HONOR Study Team. Contingency management for alcohol use disorder reduces cannabis use among American Indian and Alaska Native adults. J Subst Abuse Treat. 2022 Jun;137:108693. doi: 10.1016/j.jsat.2021.108693. Epub 2021 Dec 11. PMID 34952747
- [Derived] McDonell MG, Hirchak KA, Herron J, Lyons AJ, Alcover KC, Shaw J, Kordas G, Dirks LG, Jansen K, Avey J, Lillie K, Donovan D, McPherson SM, Dillard D, Ries R, Roll J, Buchwald D; HONOR Study Team. Effect of Incentives for Alcohol Abstinence in Partnership With 3 American Indian and Alaska Native Communities: A Randomized Clinical Trial. JAMA Psychiatry. 2021 Jun 1;78(6):599-606. doi: 10.1001/jamapsychiatry.2020.4768. PMID 33656561